CLINICAL TRIAL: NCT00896623
Title: Pharmacogenetics in Relation to Breast Cancer Outcomes in SWOG 8897
Brief Title: SWOG 8897-A DNA Analysis in Predicting Treatment Outcome in Women With Breast Cancer in SWOG 8897
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000529126; SWOG-8897-ICSC
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Amplified Fragment Length Polymorphism Analysis; Spectrometry, Mass, Matrix-Assisted Laser Desorption-Ionization

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: mutation analysis
Genetic: polymorphism analysis
Other: surface-enhanced laser desorption/ionization-time of flight mass spectrometry

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict a patient's response to treatment.

PURPOSE: This laboratory study is looking at DNA in tissue samples from women with breast cancer to see if it can predict treatment outcome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine if polymorphisms resulting in greater activation of cyclophosphamide (CYP2B6, CYP3A4, and CYP3A5) are associated with disease-free survival and treatment toxicities in women with breast cancer.
* Determine if polymorphisms resulting in less production of quinone-related oxidative damage of doxorubicin hydrochloride (NQO1, NQO2, NOS2, NOS3, CBR3) are associated with disease-free survival and treatment toxicities in these patients.

OUTLINE: This is a multicenter study.

Tissue samples archived on clinical trial SWOG-8897 are genotyped for polymorphisms in the CYP3A4, CYP3A5, CYP2B6, NQO1, NQO2, NOS2, NOS3, and CBR3 genes by matrix-assisted laser desorption ionization-time-of-flight mass spectrometry. Variant alleles are correlated with patient outcome.

PROJECTED ACCRUAL: A total of 1,577 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer

  * Node-negative breast cancer
* Enrolled on clinical trial SWOG-8897

  * Archived tissue from patients with normal lymph nodes in the low-risk group receiving no treatment and those in the intermediate group receiving treatment
* Hormone receptor status known

PATIENT CHARACTERISTICS:

* Female
* Pre- or post-menopausal

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients enrolled to SWOG 8897 consenting to banking
Sampling Method: Non-Probability Sample
Enrollment: 1577 (Actual)
Dates: Start 2006-12; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Differences in outcome according to common variant alleles | Through study follow-up an average of 10.8 years

CONTACTS AND LOCATIONS:
Overall Officials: Christine B. Ambrosone, PhD, Study Chair — Roswell Park Cancer Institute

IPD SHARING:
Plan to Share IPD: Yes
https://swog.org/Visitors/Download/Policies/Policy43.pdf

REFERENCES:
- [Result] Yao S, Barlow WE, Albain KS, Choi JY, Zhao H, Livingston RB, Davis W, Rae JM, Yeh IT, Hutchins LF, Ravdin PM, Martino S, Lyss AP, Osborne CK, Abeloff MD, Hortobagyi GN, Hayes DF, Ambrosone CB. Manganese superoxide dismutase polymorphism, treatment-related toxicity and disease-free survival in SWOG 8897 clinical trial for breast cancer. Breast Cancer Res Treat. 2010 Nov;124(2):433-9. doi: 10.1007/s10549-010-0840-0. Epub 2010 Mar 23. PMID 20309628
- [Result] Yao S, Barlow WE, Albain KS, Choi JY, Zhao H, Livingston RB, Davis W, Rae JM, Yeh IT, Hutchins LF, Ravdin PM, Martino S, Lyss AP, Osborne CK, Abeloff M, Hortobagyi GN, Hayes DF, Ambrosone CB. Gene polymorphisms in cyclophosphamide metabolism pathway,treatment-related toxicity, and disease-free survival in SWOG 8897 clinical trial for breast cancer. Clin Cancer Res. 2010 Dec 15;16(24):6169-76. doi: 10.1158/1078-0432.CCR-10-0281. PMID 21169260